CLINICAL TRIAL: NCT05496777
Title: Feasibility of Supervised Home-based Exercise Prehabilitation in Patients Scheduled for Pancreatic Resection
Brief Title: Home-based Prehabilitation in Pancreatic Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Hildebrand (Other)
Collaborators: University Medical Center Groningen (Other); University of Turin, Italy (Other)
Responsible Party: Sponsor-Investigator, Nicole Hildebrand, PhD-candidate HPB-Surgery, Academisch Ziekenhuis Maastricht
Organization: Academisch Ziekenhuis Maastricht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL75340.068.20
Record Dates: First submitted 2022-08-04; First posted 2022-08-11 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Preoperative Physical Exercise Training; Aerobic Capacity; Aerobic Fitness; Functional Mobility; Cancer; Weight, Body; Cancer of Pancreas
Keywords: Physical activity; Aerobic capacity; Body composition; Functional mobility; Pre-treatment rehabilitation; Pancreatic resection
MeSH Terms: conditions — Neoplasms; Body Weight; Pancreatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): Patients planned for pancreatic resection will be included for a home-based prehabilitation program.
  Interventions: Procedure: Home-based prehabilitation program

INTERVENTIONS:
Procedure: Home-based prehabilitation program — The home-based prehabilitation program will consist of a four-week program, where patients are expected to perform a high-intensity interval training on a home-trainer combined with functional mobility training three times a week. The program is partly supervised by a trained physiotherapist.

SUMMARY:
Rationale: The complication rate after pancreatic resection is high, especially in elderly and physically unfit patients. Aerobic capacity, as indicated by the ventilatory anaerobic threshold (VAT) assessed by a cardiopulmonary exercise test (CPET), can be used to identify high-risk patients. Previous studies have demonstrated that exercise prehabilitation can increase aerobic capacity in patients scheduled for intra-abdominal surgery, subsequently leading to better treatment outcomes. There is limited evidence on the feasibility of a (partly) supervised home-based prehabilitation program in patients scheduled for pancreatic resection.

Objective: The primary objective of this study is to assess the feasibility of a four-week supervised home-based prehabilitation program in patients scheduled for elective pancreatic resection. Secondary objectives are to evaluate individual responses to prehabilitation on a number of secondary endpoints (no cause-effect relationship to be established).

Study design: This study is a pragmatic multicenter study with a pretest-posttest design. It will take place at the Maastricht University Medical Center+ and University Medical Center Groningen in the Netherlands, and at the 'Città della Salute e della Scienza' in Torino, Italy.

Study population: Patients planned for elective resection of a pancreatic tumor will be screened for potential eligibility. High-risk patients, identified by an oxygen uptake (VO2) at VAT ≤13 ml/kg/min and/or VO2peak ≤18 ml/kg/min, will be asked to participate.

Intervention: A total of 45 patients will participate in a four-week (partly) supervised home-based personalized exercise training program before surgery (12 sessions in total). An advanced cycle ergometer (Lode Corival, Lode BV, Groningen, the Netherlands) will be delivered at the patient's home. Three weekly sessions of high-intensity interval training on the cycle will be combined with functional task exercise training. A trained physical therapist will visit the patient at least weekly to monitor progress.

Main study parameters: The main study parameter is feasibility of the (partly) supervised home-based prehabilitation program. Hereto participation rate and reasons for non-participation will be evaluated. In participating patients, adherence/compliance, dropout rate, reasons for dropout, adverse events, patient motivation, and patient and therapist appreciation will be assessed throughout the program.

Secondary endpoints: Secondary endpoints before and after prehabilitation include aerobic capacity, muscle function, body composition, functional mobility, immune system function, perceived fatigue, quality of life, and sarcopenia. Data on patient characteristics, neoadjuvant therapy, surgical procedure, and postoperative outcomes will also be collected for explorative purposes.

DETAILED DESCRIPTION:
As the aging population grows, the incidence of malignancies of the pancreas will also rise. Surgery is an important treatment modality; at the same time, it is a challenge (allostatic load) for the patient's homeostasis. Age- and disease-related psychophysiological changes and comorbidities affect tolerance to surgery (adaptive capacity). Prehabilitation may increase a patient's ability to cope with surgical-induced allostatic load by improving the capacity and functioning of the respiratory, cardiovascular, and/or musculoskeletal systems, and therefore lower the risk of postoperative morbidity and mortality.

About 28% of patients undergoing pancreatic resection developed a major complication (Clavien-Dindo grade III or higher), and 3.2% deceased in-hospital in the Netherlands between 2014 and 2017. Older patients, especially physically unfit patients, are more prone to complications.

Preoperative aerobic capacity has been found to have a consistent relationship with postoperative outcome in major elective intra-abdominal surgery, such as pancreatic resection. Previous studies consistently indicated that an oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT) <11mL/kg/min and/or a VO2 at peak exercise (VO2peak) <18mL/kg/min, as determined during a cardiopulmonary exercise test (CPET), are cut-off points to identify patients that have a higher risk for postoperative morbidity and mortality. Exercise prehabilitation has been reported to be able to preoperatively increase the physical fitness of patients scheduled for elective intra-abdominal surgery, of which high-risk patients will benefit the most. Most prehabilitation programs were carried out under supervision in an outpatient clinic. Often however, patients are not able or willing to participate, for example because of travelling issues or because it is becoming 'too much'. Home-based programs are often unsupervised and lack the ability to monitor adherence of the patient, and therefore might lack effectiveness.

A personalized exercise program in a home-based setting might enhance the participation rate, motivation, and adherence of patients. This has proven to be the preferred method for previous prehabilitation programs. Although several studies investigated the effects of exercise prehabilitation before pancreatic resection and reported positive effects on preoperative physical fitness and postoperative morbidity, there is limited evidence addressing the feasibility and effectiveness of (partly) supervised home-based prehabilitation in these populations. Moreover, effectiveness has not been evaluated using sophisticated outcome measures.

In a recent study in patients planned for liver or pancreatic surgery the adherence rate of a semi-supervised home-based training program was 83%. Furthermore, it led to an increase in VO2 at the VAT of 17.8% and VO2peak of 17.2%. This leads to the hypothesis that a partly supervised home-based prehabilitation program is feasible in a high risk-group. To test this hypothesis further the study will investigate the feasibility of a (partly) supervised prehabilitation program and will focus on patients undergoing pancreatic resection.

Objectives:

The primary objective of the study is to assess feasibility of a four-week (partly) supervised home-based prehabilitation program in patients scheduled for elective pancreatic resection. This will be measured using participation rate, reasons for non-participation, adherence/compliance, dropout rate, reasons for dropout, adverse events, patient motivation, and patient and therapist appreciation.

Secondary objectives are to evaluate individual responses to prehabilitation on the secondary study parameters. Data on patient characteristics, neoadjuvant therapy, surgical procedure, and postoperative outcomes will also be collected for explorative purposes.

Study design:

This study is a pragmatic multicenter study with a pretest-posttest design. It will take place at the Maastricht University Medical Center+ and University Medical Center Groningen in the Netherlands, as well as at the 'Città della Salute e della Scienza' in Torino, Italy.

Patients planned for elective pancreatic resection will be screened for CPET by a trained oncology nurse specialist. A trained medical physiologist will perform the CPET. Patients are eligible for the study if they have an oxygen uptake (VO2) at the VAT of ≤13 ml/kg/min and/or VO2peak ≤18 ml/kg/min. Potential candidates will be given full details of the study and invited to participate. If patients give permission, they will be contacted by an investigator who provides extensive information about the study.

If patients sign informed consent, they will fill out the baseline questionnaires (perceived fatigue, quality of life, and sarcopenia), and undergo baseline testing. Baseline tests include body composition, functional mobility, questionnaires, and immune system function.

After baseline assessment an advanced cycle ergometer (Lode Corival Home+, Lode BV, Groningen, the Netherlands) will be delivered to the patient's home. A trained community physical therapist will visit the patient at home to explain correct use of the ergometer and to (partly) supervise training program. A steep ramp test will be carried out by the physical therapist. The high-intensity interval exercise training program on the cycle ergometer will be personalized based on a weekly supervised steep ramp test. Every training session on the ergometer will take 30 minutes. Next to training at the cycle ergometer, patients will complete 15 minutes of functional exercises (e.g., sit-to-stand exercises, stair-climbing, cycling, walking). The patient will be asked to perform different types of exercises, a total of 15 exercises of about 30 seconds, with 30 seconds of rest in between. The physical therapist will explain the functional exercises and supervise the patient in the first week. Based on the patient's progress in muscle function and functional mobility, which will be tested weekly using the 30-second chair stand test at the patient's home, the physical therapist will adjust the exercises weekly. Patients will be asked to train three times a week for four weeks. In the first week, the physical therapist visits three times, whereas the patient will be visited once a week in week 2, 3, and 4.

After the prehabilitation program, patient and therapist will fill out an appreciation questionnaire. The other questionnaires will be filled in again. Also, tests on aerobic capacity, body composition, functional mobility, and immune system function will be repeated.

Aerobic capacity A maximal CPET will be performed using a calibrated electronically braked cycle. Patients with contraindications for CPET due to cardiorespiratory comorbidities will not be able to participate in the study. The patient will be fitted with an electrocardiogram, as well as a calibrated respiratory gas analysis system, that will calculate breath-by-breath VO2, carbon dioxide production (VCO2), and minute ventilation. Blood pressure and peripheral oxygen saturation will be monitored. After two minutes of rest measurements, the patient starts cycling unloaded for 2 minutes. Thereafter, depending on the patient's physical fitness, the work rate will be linearly incremented with a 5, 10, 15, or 20W/min ramp protocol to ensure a test duration between eight and twelve minutes. Patients will be instructed to maintain a pedaling frequency of 80/min. Test effort will be considered maximal when the patient shows objective (heart rate at peak exercise >95% of predicted and/or a respiratory exchange ratio at peak exercise >1.10) and subjective (unsteady biking, sweating, facial flushing, inability to continue despite encouragement) signs of maximal effort. Perceived exertion before and directly after CPET, using a ten-point visual analog scale, will be asked. CPET interpretation will be performed by a trained and experienced medical physiologist. The ventilatory anaerobic threshold is defined as the point at which the ventilatory equivalent for oxygen and the partial end-tidal oxygen tension reached a minimum and thereafter began to rise in a consistent manner, coinciding with an unchanged ventilatory equivalent for carbon dioxide and partial end-tidal carbon dioxide tension. If this method appeared to provide uncertain results, the V-slope method will be used.

A steep ramp test will be performed on a weekly base at the patient's home under supervision of a physical therapist to assess and monitor aerobic fitness. The advanced cycle ergometer will be used for the steep ramp test. The patient will be fitted a heart rate belt around the chest (Polar Elektro Oy, Kempele, Finland) during the test. After three minutes of rest the test will start and the work rate will be increased by a constant increment of 10 W every 10 seconds in a ramp like manner. Test duration will be four to seven minutes. The pedaling frequency should be kept constant between 60 and 80 revolutions per minute. Peak exercise is the point at which there is a sustained drop in pedaling frequency from 60 revolutions per minute, despite verbal encouragement. Data will be stored for further use. A ten-point VAS will be used to ask the level of perceived exertion. The attained peak work rate (WRpeak) will be used to adjust the training protocol for the upcoming week.

Muscle function Muscle function measurement will be measured for patients in Città della Salute e della Scienza. Knee extensors torque will be recorded using an isokinetic device under isometric sub-maximal and maximal voluntary contractions. The rate of torque development will be calculated for each contraction at different submaximal amplitudes (from 20% to 80% of maximal voluntary torque). Lastly, to measure muscle fatigability, participants will perform a submaximal isometric contraction at 70% of maximal voluntary torque until task failure (the time failure typically occurs within 60 s). High-density surface electromyographic (HDEMG) signals will be recorded from the vastus lateralis and medialis muscle during all muscle contractions to record muscle fiber conduction velocity. Muscle fiber conduction velocity is an important physiological variable associated to the qualities of skeletal muscles. Furthermore, HDEMG signals will be decomposed to identify and assess the activity of a large number of motor units over a wide range of torques, providing direct evidence on the strategies used by the central nervous system to control muscle torque.

Body composition The patient's body mass and body height will be measured pre-, and post-intervention. Body mass will be measured weekly at the patient's home. To assess skeletal muscle mass and quality a single slice of the patient's abdominal CT-scan will be selected at the level of the third lumbar vertebra (L3). Scans will be analyzed using an automated segmentation system developed and validated at Maastricht University. Skeletal muscle, visceral adipose tissue, and subcutaneous adipose tissue areas will be normalized for the patient's body height to calculate the L3 index in cm2/m2. Skeletal muscle radiation attenuation will be assessed by calculating the average Hounsfield Units value of skeletal muscle mass.

Functional mobility Functional mobility will be assessed in all patients using the 30-second chair-stand test pre- and post-intervention at the hospital, and weekly at the patient's home. Additionally, a 2-minute walk test will be performed pre- and post-intervention. The 30-second chair-stand test evaluates a combination of functional mobility, balance, and lower leg muscle strength. The primary outcome is the repetitions of standing up from a sitting position and sitting back down with crossed arms within 30 seconds. The 2-minute walk test records the distance in meters that is walked within two minutes, with a walking aid if necessary.

Immunological phenotyping Given the evidence that exercise leads to changes in the innate and adaptive immune system, blood samples will be drawn pre- and post-intervention. Levels of interleukin 6, interleukin 8, and interleukin 10, as well as C-reactive protein, and tumor necrosis factor-α will be measured by multiplex analysis. Blood samples will be centrifuged, and plasma will be stored in aliquots at -80 °C until assayed for future analysis. Blood samples will be stored, for a maximum of ten years, in the biobank of the participating hospital. Future analysis must be in line with the aims of our current research; if not, informed consent must be obtained.

Questionnaires Patients will fill out the multidimensional fatigue index, a self-reporting questionnaire with 20 propositions about different dimensions and consequences of fatigue. A higher score means a higher level of perceived fatigue. Patients will also fill out the European Organisation for Research and Treatment of Cancer Quality of Life questionnaire (EORTC QLQ-C30), a questionnaire with 30 items in four domains developed to assess the quality of life in cancer patients. A difference to baseline of 10 points can be considered clinically relevant. The SARC-F, a five-item questionnaire on the consequences of sarcopenia will also be filled out by the patients.

Preoperative patient characteristics:

Relevant demographic data (e.g., age and sex of participants), diagnosis, American Society of Anesthesiologists score, and Charlson comorbidity index will be collected preoperatively.

Postoperative care Details on type of surgery and intraoperative outcomes will also be collected. According to standard of care, all patients will receive postoperative physical therapy after surgery in all three participating centers. Postoperative complications will be recorded for 30 days and scored according to the Clavien-Dindo classification. The 30-day readmission rate will also be recorded. Surgical outcomes will be obtained from the electronic patient record system and from patient's physical examination on the ward.

ELIGIBILITY:
Inclusion Criteria:

* An oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT) ≤13 ml/kg/min and/or an VO2peak ≤18 ml/kg/min assessed using cardiopulmonary exercise testing
* Age ≥18 years
* Scheduled for elective pancreatic resection at Maastricht UMC+, at the University Medical Center Groningen, or the Citta della Salute e della Scienza Hospital in Torino
* Willing to participate in the home-based prehabilitation program
* Providing informed consent to participate

Exclusion Criteria:

* Patients requiring acute (emergency) surgery;
* Patients undergoing surgery in another hospital;
* Patients not living within the catchment area of the hospital (<30 minutes);
* Patients not capable of cycling on a cycle ergometer;
* Patients with contraindications for physical exercise training;
* Unable to cooperate with the testing procedures (e.g., insufficient understanding of the Dutch or Italian language at the Maastricht University Medical Center+, at the University Medical Center Groningen, or at the 'Città della Salute e della Scienza' Hospital in Torino, respectively);
* No physical therapist with the right education (functional task training/home based prehabilitation) available in the living area of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Participation rate | At recruitment
  Rate of eligible patients that participate in the prehabilitation program
Reasons for non-participation | At recruitment
  Patient's reasons for non-participation in the prehabilitation program while being eligible
Adherence/compliance | 4-week training period
  Adherence rate to the prehabilitation program
Dropout rate | 4-week training period
  Dropout rate of the prehabilitation program
Reasons for dropout | 4-week training period, at moment of drop-out
  Participant's reasons for dropping out the prehabilitation program
Adverse events | 4-week training period
  Any undesirable experience occurring to a participant during the study, whether or not considered related to the experimental supervised home-based prehabilitation program
Patient appreciation | at the end of 4-week training period
  Patient appreciation measured via an appreciation questionnaire
Therapist appreciation | at the end of 4-week training period
  Therapist appreciation measured via an appreciation questionnaire

SECONDARY OUTCOMES:
Aerobic capacity | 4 weeks (pre- and post-prehabiltation)
  Oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT) and VO2peak
Muscle function | 4 weeks (pre- and post-prehabiltation)
  Knee extensors torque in an isokinetic device under isometric submaximal and maximal voluntary contractions
Body composition | 4 weeks (pre- and post-prehabiltation)
  Automated segmentation of body composition on L3 level of abdominal CT-scans
Functional mobility/muscle strength | 4 weeks (pre- and post-prehabiltation)
  2-minute walk test
Functional mobility/muscle strength | Weekly during 4-week training period
  30-second chair-stand test
Immune system function | 4 weeks (pre- and post-prehabiltation)
  Immunological phenotyping
Level of perceived fatigue | 4 weeks (pre- and post-prehabiltation)
  Multidimensional fatigue index
Quality of life measurement | 4 weeks (pre- and post-prehabiltation)
  European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Olde Damink, M.D., M.Sc., PhD, Principal Investigator — Maastricht University Medical Center
Locations (3):
- Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino, Italy
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center+, Maastricht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bongers BC, Dejong CHC, den Dulk M. Enhanced recovery after surgery programmes in older patients undergoing hepatopancreatobiliary surgery: what benefits might prehabilitation have? Eur J Surg Oncol. 2021 Mar;47(3 Pt A):551-559. doi: 10.1016/j.ejso.2020.03.211. Epub 2020 Mar 29. PMID 32253075
- [Background] Ngo-Huang A, Parker NH, Wang X, Petzel MQB, Fogelman D, Schadler KL, Bruera E, Fleming JB, Lee JE, Katz MHG. Home-based exercise during preoperative therapy for pancreatic cancer. Langenbecks Arch Surg. 2017 Dec;402(8):1175-1185. doi: 10.1007/s00423-017-1599-0. Epub 2017 Jul 15. PMID 28710540
- [Background] Ferreira V, Agnihotram RV, Bergdahl A, van Rooijen SJ, Awasthi R, Carli F, Scheede-Bergdahl C. Maximizing patient adherence to prehabilitation: what do the patients say? Support Care Cancer. 2018 Aug;26(8):2717-2723. doi: 10.1007/s00520-018-4109-1. Epub 2018 Feb 24. PMID 29478189
- [Background] Driessen EJ, Peeters ME, Bongers BC, Maas HA, Bootsma GP, van Meeteren NL, Janssen-Heijnen ML. Effects of prehabilitation and rehabilitation including a home-based component on physical fitness, adherence, treatment tolerance, and recovery in patients with non-small cell lung cancer: A systematic review. Crit Rev Oncol Hematol. 2017 Jun;114:63-76. doi: 10.1016/j.critrevonc.2017.03.031. Epub 2017 Apr 5. PMID 28477748
- [Background] Parker NH, Lee RE, O'Connor DP, Ngo-Huang A, Petzel MQB, Schadler K, Wang X, Xiao L, Fogelman D, Simpson R, Fleming JB, Lee JE, Tzeng CD, Sahai SK, Basen-Engquist K, Katz MHG. Supports and Barriers to Home-Based Physical Activity During Preoperative Treatment of Pancreatic Cancer: A Mixed-Methods Study. J Phys Act Health. 2019 Dec 1;16(12):1113-1122. doi: 10.1123/jpah.2019-0027. Epub 2019 Oct 7. PMID 31592772
- [Background] van Wijk L, Bongers BC, Berkel AEM, Buis CI, Reudink M, Liem MSL, Slooter GD, van Meeteren NLU, Klaase JM. Improved preoperative aerobic fitness following a home-based bimodal prehabilitation programme in high-risk patients scheduled for liver or pancreatic resection. Br J Surg. 2022 Oct 14;109(11):1036-1039. doi: 10.1093/bjs/znac230. No abstract available. PMID 35851601
- [Background] Hulzebos EH, van Meeteren NL. Making the elderly fit for surgery. Br J Surg. 2016 Mar;103(4):463. doi: 10.1002/bjs.10134. No abstract available. PMID 26891214
- [Background] van Roessel S, Mackay TM, van Dieren S, van der Schelling GP, Nieuwenhuijs VB, Bosscha K, van der Harst E, van Dam RM, Liem MSL, Festen S, Stommel MWJ, Roos D, Wit F, Molenaar IQ, de Meijer VE, Kazemier G, de Hingh IHJT, van Santvoort HC, Bonsing BA, Busch OR, Groot Koerkamp B, Besselink MG; Dutch Pancreatic Cancer Group. Textbook Outcome: Nationwide Analysis of a Novel Quality Measure in Pancreatic Surgery. Ann Surg. 2020 Jan;271(1):155-162. doi: 10.1097/SLA.0000000000003451. PMID 31274651
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Wilson RJ, Davies S, Yates D, Redman J, Stone M. Impaired functional capacity is associated with all-cause mortality after major elective intra-abdominal surgery. Br J Anaesth. 2010 Sep;105(3):297-303. doi: 10.1093/bja/aeq128. Epub 2010 Jun 23. PMID 20573634
- [Background] Moran J, Wilson F, Guinan E, McCormick P, Hussey J, Moriarty J. Role of cardiopulmonary exercise testing as a risk-assessment method in patients undergoing intra-abdominal surgery: a systematic review. Br J Anaesth. 2016 Feb;116(2):177-91. doi: 10.1093/bja/aev454. PMID 26787788
- [Background] Smith TB, Stonell C, Purkayastha S, Paraskevas P. Cardiopulmonary exercise testing as a risk assessment method in non cardio-pulmonary surgery: a systematic review. Anaesthesia. 2009 Aug;64(8):883-93. doi: 10.1111/j.1365-2044.2009.05983.x. PMID 19604193
- [Background] Hightower CE, Riedel BJ, Feig BW, Morris GS, Ensor JE Jr, Woodruff VD, Daley-Norman MD, Sun XG. A pilot study evaluating predictors of postoperative outcomes after major abdominal surgery: Physiological capacity compared with the ASA physical status classification system. Br J Anaesth. 2010 Apr;104(4):465-71. doi: 10.1093/bja/aeq034. Epub 2010 Feb 26. PMID 20190255
- [Background] Hartley RA, Pichel AC, Grant SW, Hickey GL, Lancaster PS, Wisely NA, McCollum CN, Atkinson D. Preoperative cardiopulmonary exercise testing and risk of early mortality following abdominal aortic aneurysm repair. Br J Surg. 2012 Nov;99(11):1539-46. doi: 10.1002/bjs.8896. Epub 2012 Sep 21. PMID 23001820
- [Background] Prentis JM, Trenell MI, Jones DJ, Lees T, Clarke M, Snowden CP. Submaximal exercise testing predicts perioperative hospitalization after aortic aneurysm repair. J Vasc Surg. 2012 Dec;56(6):1564-70. doi: 10.1016/j.jvs.2012.05.097. Epub 2012 Aug 2. PMID 22858436
- [Background] Prentis JM, Manas DM, Trenell MI, Hudson M, Jones DJ, Snowden CP. Submaximal cardiopulmonary exercise testing predicts 90-day survival after liver transplantation. Liver Transpl. 2012 Feb;18(2):152-9. doi: 10.1002/lt.22426. PMID 21898768
- [Background] Chandrabalan VV, McMillan DC, Carter R, Kinsella J, McKay CJ, Carter CR, Dickson EJ. Pre-operative cardiopulmonary exercise testing predicts adverse post-operative events and non-progression to adjuvant therapy after major pancreatic surgery. HPB (Oxford). 2013 Nov;15(11):899-907. doi: 10.1111/hpb.12060. Epub 2013 Feb 20. PMID 23458160
- [Background] West MA, Asher R, Browning M, Minto G, Swart M, Richardson K, McGarrity L, Jack S, Grocott MP; Perioperative Exercise Testing and Training Society. Validation of preoperative cardiopulmonary exercise testing-derived variables to predict in-hospital morbidity after major colorectal surgery. Br J Surg. 2016 May;103(6):744-752. doi: 10.1002/bjs.10112. Epub 2016 Feb 23. PMID 26914526
- [Background] Junejo MA, Mason JM, Sheen AJ, Bryan A, Moore J, Foster P, Atkinson D, Parker MJ, Siriwardena AK. Cardiopulmonary exercise testing for preoperative risk assessment before pancreaticoduodenectomy for cancer. Ann Surg Oncol. 2014 Jun;21(6):1929-36. doi: 10.1245/s10434-014-3493-0. Epub 2014 Jan 30. PMID 24477709
- [Background] Ausania F, Snowden CP, Prentis JM, Holmes LR, Jaques BC, White SA, French JJ, Manas DM, Charnley RM. Effects of low cardiopulmonary reserve on pancreatic leak following pancreaticoduodenectomy. Br J Surg. 2012 Sep;99(9):1290-4. doi: 10.1002/bjs.8859. Epub 2012 Jul 24. PMID 22828960
- [Background] Older P, Smith R, Courtney P, Hone R. Preoperative evaluation of cardiac failure and ischemia in elderly patients by cardiopulmonary exercise testing. Chest. 1993 Sep;104(3):701-4. doi: 10.1378/chest.104.3.701. PMID 8365279
- [Background] Bruns ER, van den Heuvel B, Buskens CJ, van Duijvendijk P, Festen S, Wassenaar EB, van der Zaag ES, Bemelman WA, van Munster BC. The effects of physical prehabilitation in elderly patients undergoing colorectal surgery: a systematic review. Colorectal Dis. 2016 Aug;18(8):O267-77. doi: 10.1111/codi.13429. PMID 27332897
- [Background] Thomas G, Tahir MR, Bongers BC, Kallen VL, Slooter GD, van Meeteren NL. Prehabilitation before major intra-abdominal cancer surgery: A systematic review of randomised controlled trials. Eur J Anaesthesiol. 2019 Dec;36(12):933-945. doi: 10.1097/EJA.0000000000001030. PMID 31188152
- [Background] Dunne DF, Jack S, Jones RP, Jones L, Lythgoe DT, Malik HZ, Poston GJ, Palmer DH, Fenwick SW. Randomized clinical trial of prehabilitation before planned liver resection. Br J Surg. 2016 Apr;103(5):504-12. doi: 10.1002/bjs.10096. Epub 2016 Feb 11. PMID 26864728
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Nakajima H, Yokoyama Y, Inoue T, Nagaya M, Mizuno Y, Kadono I, Nishiwaki K, Nishida Y, Nagino M. Clinical Benefit of Preoperative Exercise and Nutritional Therapy for Patients Undergoing Hepato-Pancreato-Biliary Surgeries for Malignancy. Ann Surg Oncol. 2019 Jan;26(1):264-272. doi: 10.1245/s10434-018-6943-2. Epub 2018 Oct 26. PMID 30367303
- [Background] Lundberg M, Archer KR, Larsson C, Rydwik E. Prehabilitation: The Emperor's New Clothes or a New Arena for Physical Therapists? Phys Ther. 2019 Feb 1;99(2):127-130. doi: 10.1093/ptj/pzy133. No abstract available. PMID 30508203
- [Background] Ngo-Huang A, Parker NH, Bruera E, Lee RE, Simpson R, O'Connor DP, Petzel MQB, Fontillas RC, Schadler K, Xiao L, Wang X, Fogelman D, Sahai SK, Lee JE, Basen-Engquist K, Katz MHG. Home-Based Exercise Prehabilitation During Preoperative Treatment for Pancreatic Cancer Is Associated With Improvement in Physical Function and Quality of Life. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419894061. doi: 10.1177/1534735419894061. PMID 31858837
- [Background] Parker NH, Ngo-Huang A, Lee RE, O'Connor DP, Basen-Engquist KM, Petzel MQB, Wang X, Xiao L, Fogelman DR, Schadler KL, Simpson RJ, Fleming JB, Lee JE, Varadhachary GR, Sahai SK, Katz MHG. Physical activity and exercise during preoperative pancreatic cancer treatment. Support Care Cancer. 2019 Jun;27(6):2275-2284. doi: 10.1007/s00520-018-4493-6. Epub 2018 Oct 17. PMID 30334105
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Courneya KS. Exercise interventions during cancer treatment: biopsychosocial outcomes. Exerc Sport Sci Rev. 2001 Apr;29(2):60-4. doi: 10.1097/00003677-200104000-00004. PMID 11337824
- [Background] Hjermstad MJ, Fossa SD, Bjordal K, Kaasa S. Test/retest study of the European Organization for Research and Treatment of Cancer Core Quality-of-Life Questionnaire. J Clin Oncol. 1995 May;13(5):1249-54. doi: 10.1200/JCO.1995.13.5.1249. PMID 7738629
- [Background] Nguyen TN, Nguyen AT, Khuong LQ, Nguyen TX, Nguyen HTT, Nguyen TTH, Hoang MV, Pham T, Nguyen TN, Vu HTT. Reliability and Validity of SARC-F Questionnaire to Assess Sarcopenia Among Vietnamese Geriatric Patients. Clin Interv Aging. 2020 Jun 9;15:879-886. doi: 10.2147/CIA.S254397. eCollection 2020. PMID 32606628
- [Background] Cuijpers ACM, Heldens AFJM, Bours MJL, van Meeteren NLU, Stassen LPS, Lubbers T, Bongers BC. Relation between preoperative aerobic fitness estimated by steep ramp test performance and postoperative morbidity in colorectal cancer surgery: prospective observational study. Br J Surg. 2022 Feb 1;109(2):155-159. doi: 10.1093/bjs/znab292. PMID 34536001
- [Background] Lamarra N, Whipp BJ, Ward SA, Wasserman K. Effect of interbreath fluctuations on characterizing exercise gas exchange kinetics. J Appl Physiol (1985). 1987 May;62(5):2003-12. doi: 10.1152/jappl.1987.62.5.2003. PMID 3110126
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Ackermans LLGC, Volmer L, Wee L, Brecheisen R, Sanchez-Gonzalez P, Seiffert AP, Gomez EJ, Dekker A, Ten Bosch JA, Olde Damink SMW, Blokhuis TJ. Deep Learning Automated Segmentation for Muscle and Adipose Tissue from Abdominal Computed Tomography in Polytrauma Patients. Sensors (Basel). 2021 Mar 16;21(6):2083. doi: 10.3390/s21062083. PMID 33809710
- [Background] Taaffe DR, Henwood TR, Nalls MA, Walker DG, Lang TF, Harris TB. Alterations in muscle attenuation following detraining and retraining in resistance-trained older adults. Gerontology. 2009;55(2):217-23. doi: 10.1159/000182084. Epub 2008 Dec 5. PMID 19060453
- [Background] Snyder CF, Blackford AL, Sussman J, Bainbridge D, Howell D, Seow HY, Carducci MA, Wu AW. Identifying changes in scores on the EORTC-QLQ-C30 representing a change in patients' supportive care needs. Qual Life Res. 2015 May;24(5):1207-16. doi: 10.1007/s11136-014-0853-y. Epub 2014 Nov 15. PMID 25398495
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Derived] Hildebrand ND, Wijma AG, Bongers BC, Rensen SS, den Dulk M, Klaase JM, Olde Damink SWM. Adherence and response to supervised home-based exercise prehabilitation of unfit patients scheduled for pancreatic surgery. Eur J Surg Oncol. 2025 Oct;51(10):110302. doi: 10.1016/j.ejso.2025.110302. Epub 2025 Jul 4. PMID 40652824
- [Derived] Hildebrand ND, Wijma AG, Bongers BC, Rensen SS, den Dulk M, Klaase JM, Olde Damink SWM. Supervised Home-Based Exercise Prehabilitation in Unfit Patients Scheduled for Pancreatic Surgery: Protocol for a Multicenter Feasibility Study. JMIR Res Protoc. 2023 Sep 7;12:e46526. doi: 10.2196/46526. PMID 37676715